CLINICAL TRIAL: NCT03874169
Title: Detection of Gastrointestinal Bleeding in Intensive Care Patients Via Biosensor Watch
Status: Terminated | Type: Observational
Why Stopped: Due to the COVID-19 Pandemic
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAS1510
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Gastro Intestinal Bleeding
Keywords: Biosensor watch; E4 Wristband; Intensive Care Unit; GI bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- High-Risk of GI Bleed: Patients that have a high risk of having a gastrointestinal bleed upon admission into the ICU based on their medical history and symptoms. These patients will have a biosensor watch, the E4 wristband, placed on them to monitor their vital signs.
  Interventions: Device: E4 wristband

INTERVENTIONS:
Device: E4 wristband — A biosensor watch that monitors the patient's heartbeat, heart rate variability, skin conductance, and temperature in order to discover if they are having a GI bleed

SUMMARY:
The purpose of this study to improve methods of monitoring and diagnosing gastrointestinal bleeding via the E4 wristband, a biosensor watch.

DETAILED DESCRIPTION:
The annual occurrence of gastrointestinal (GI) bleeding is approximately 150 per 100,000 in the US and accounts for 300,000 hospitalizations per year with a death rate of 5%. Qualitative assessments of blood tests monitoring patients with or are thought to have GI bleeding can lack accuracy and objectivity, delaying conformation of the bleed through endoscopy. Early endoscopies have been linked to more favorable outcomes for patients with heavier GI bleeding and earlier discharge times for patients with less severe GI bleeding. Additionally, laboratory values are not documented at regular intervals, which makes identifying when GI bleeding exactly occurred difficult. In this study, the investigators aim to improve methods of monitoring and diagnosing GI bleeding via the E4 wristband, a biosensor watch. Using data from the E4 wristband, the investigators will train a model to recognize GI bleeding through analyzing the heart rate and skin conductance of both patients with GI bleeding and who may have GI bleeding while they are not bleeding and while they are bleeding. Monitoring both types of patients while they are and are not bleeding will help the model discern which vital signs are critical. Additionally, the investigators will be using blood tests and other traditional methods of diagnosis to create a standard for vitals that characterize GI bleeding. If the E4 wristband is successfully able to accurately identify when a patient is experiencing GI bleeding, then speed of GI bleeding detection and the ability to monitor GI bleeding will dramatically increase, leading to quicker discharge times, reduced risk of rebleeding, and a lower death rate for afflicted patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of gastrointestinal bleeding and/or showing the symptoms of gastrointestinal bleeding.

Exclusion Criteria:

* Patients who are not showing the symptoms of gastrointestinal bleeding and/or do not have a history of gastrointestinal bleeding.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the intensive care unit (ICU) in the Milstein Hospital Building at Columbia University.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Heart Rate | Up to 1 year
  Using the wristband, heart rate will be collected at a frequency of 64 Hz.
Skin Conductance | Up to 1 year
  Using the wristband, skin conductance will be collected at a frequency of 4 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Chin Hur, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share with other researchers outside of the research team.

REFERENCES:
- [Background] Kim BS, Li BT, Engel A, Samra JS, Clarke S, Norton ID, Li AE. Diagnosis of gastrointestinal bleeding: A practical guide for clinicians. World J Gastrointest Pathophysiol. 2014 Nov 15;5(4):467-78. doi: 10.4291/wjgp.v5.i4.467. PMID 25400991